CLINICAL TRIAL: NCT03614299
Title: Pateint-reported Outcomes and Objective Eye Dryness Evaluation in Primary Sjögren's Syndrome.
Brief Title: Eye Dryness Evaluation in Primary Sjögren's Syndrome
Acronym: PEPSS
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC18.0173
Record Dates: First submitted 2018-07-31; First posted 2018-08-03 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Primary Sjögren Syndrome
MeSH Terms: interventions — Microscopy, Interference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, saliva, cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pSS cohort: Patients with pSS included in the study
  Interventions: Other: Ecological symptom measurements using a webapp; Diagnostic Test: Interferometry

INTERVENTIONS:
Other: Ecological symptom measurements using a webapp — A webapp will be installed on the patients' smartphone, which will be used to collect everyday the symptoms of the patients (ESSPRI score)
Diagnostic Test: Interferometry — Evaluation of the mebomian function using the LipiView methodology

SUMMARY:
The objective of this observational study is to develop new tools to assess primary Sjögren's syndrome (pSS) symptoms and to measure the severity of eye involvement in these patients.

DETAILED DESCRIPTION:
All clinical trials evaluating the efficacy of immunomodulatory drugs in pSS are negative. This could be due to a lack of sensitivity of the outcome measures used so far to define the response. In this study, investigator will evaluate the feasability, tolerability, and performance of new tools to assess disease evolution:

* investigator will develop a webapp to measure the intensity of the symptoms at home on a daily basis (ecological assessment)
* investigator will evaluate new ophthalmologic procedures, already used in other conditions but never in pSS, which assess the severity of eye involvement in the disease
* investigator will develop an automated method to score the severity of ocular surface lesions in the disease.

Patients with a diagnosis of pSS will be included in the study, will undergo detailed ophtalmologic examination, and will then use a webapp, installed on their smartphone, to score their symptoms everyday during 3 months.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of pSS according to ACR/EULAR classification criteria

Exclusion Criteria:

* patient does not possess a smartphone with web connection
* patient unable to sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive pSS patients seen in Rheumatology
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Variability in the intensity of patient-reported symptoms | 3 months
  Variability over time (day-to-day assessment) of the ESSPRI score (dispersion of the values compared to the mean)

SECONDARY OUTCOMES:
Tolerability of the daily use of a webapp to measure the symptoms | Month 3
  Score Questionnaire SUS - System Usability Scale. The SUS ranges from 0 to 100, with values above 68 considered as above average.
Interferometry | 3 months
  Measure of mebomian function using the LipiView technology
Automated eye surface coloration measurement | 3 months
  Development of an automated method using deep image mining on recorded videos

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de BREST, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning after publication of result and ending three years maximum following the last visit of last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.